CLINICAL TRIAL: NCT05907304
Title: An Open-label Study to Assess the Safety and Efficacy of Naporafenib (ERAS-254) Administered With Trametinib in Previously Treated Patients With Locally Advanced Unresectable or Metastatic Solid Tumor Malignancies With RAS Q61X Mutations
Brief Title: A Study to Assess Naporafenib (ERAS-254) Administered With Trametinib in Patients With RAS Q61X Mutations
Acronym: SEACRAFT-1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Erasca, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERAS-254-01
Record Dates: First submitted 2023-05-30; First posted 2023-06-18 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: Melanoma; Non-small cell lung cancer; Thyroid cancer; Colorectal Cancer (cohort full); Pancreatic Cancer; Other solid tumors harboring a RAS Q61X mutation
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Thyroid Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms | interventions — naporafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Naporafenib + Trametinib (Experimental): Naporafenib (ERAS-254) 200 mg twice daily (BID) Trametinib 1 mg once daily (QD)
  Interventions: Drug: Naporafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Naporafenib — Naporafenib (ERAS-254) 200 mg twice daily (BID) of an experimental Pan-Raf inhibitor
  Other Names: LXH254; ERAS-254
Drug: Trametinib — Trametinib is an FDA approved anticancer medication that targets MEK1 and MEK2.
  Other Names: Mekinist

SUMMARY:
To evaluate the efficacy of naporafenib administered with trametinib in patients with rat sarcoma viral oncogene (RAS) Q61X solid tumors

* To evaluate the safety and tolerability of naporafenib administered with trametinib in patients with RAS Q61X solid tumors
* To characterize the pharmacokinetic (PK) profile of naporafenib and trametinib when administered to patients with RAS Q61X solid tumors

DETAILED DESCRIPTION:
SEACRAFT-1 is an open-label study to assess the safety and efficacy of naporafenib administered with trametinib in previously treated patients with locally advanced unresectable or metastatic RAS Q61X solid tumor malignancies. The study will enroll a total of approximately 100 adult patients; a sub-study will enroll approximately 15 adolescent patients ≥12 and <18 years for a total sample size of approximately 115. Patients with a locally advanced unresectable or metastatic solid tumor malignancy that is not responsive to standard therapies or for which there is no standard therapy are eligible. Patients with primary central nervous system (CNS) tumors are not eligible. Documentation of a RAS Q61X mutation in tumor tissue prior to the first dose of study treatment is required.

ELIGIBILITY:
Key Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Age ≥ 12 years
3. A locally advanced or metastatic tumor who has progressed on or for which no standard therapy exists. Patients who are intolerant to standard therapy or who are not a candidate for standard therapy (in the opinion of the Investigator) or who decline standard therapy are also eligible.
4. Documentation of a RAS Q61X mutation (tumor tissue or blood) prior to first dose of study treatment as determined locally with an analytically validated assay in a certified testing laboratory.
5. Archival tumor tissue collected within 5 years prior to enrollment must be confirmed to be available at the time of Screening, which may be submitted before or after enrollment for exploratory biomarker analysis.
6. ECOG performance status 0, 1 or 2
7. Presence of at least 1 measurable lesion according to RECIST v1.1
8. Able to swallow oral medication.

Exclusion Criteria:

1. Prior therapy with an ERK-, MEK-, RAF-, or RAS-inhibitor
2. Impairment of GI function or gastrointestinal (GI) disease that may significantly alter the absorption of study treatment (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection)
3. History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndrome)
4. Corrected QT interval using Fridericia's formula (QTcF) at Screening >450 ms based on triplicate average NOTE: criterion does not apply to patients with a right or left bundle branch block
5. LVEF <50%
6. All primary CNS tumors
7. Symptomatic CNS metastases that are neurologically unstable. Patients with controlled CNS metastases are eligible.
8. Patients receiving treatment with medications that are known to be strong inhibitors and/or inducers of cytochrome P450 (CYP)3A; substrates of CYP2C8, CYP2C9, and CYP3A with a narrow therapeutic index and sensitive substrates of CYP3A;
9. Are pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of naporafenib administered with trametinib in patients with rat sarcoma viral oncogene (RAS) Q61X solid tumors | Assessed up to 24 months from time of first dose
  Based on assessment of Objective response rate (ORR) per RECIST version 1.1

SECONDARY OUTCOMES:
Adverse Events | Assessed up to 24 months from time of first dose
  Incidence and severity of treatment-emergent AEs and serious AEs
Duration of Response (DOR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1
Time to Response (TTR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1
Progression Free Survival (PFS) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1
Disease Control Rate (DCR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1
Plasma concentration (Cmax) | Study Day 1 up to Day 29
  Maximum plasma concentration of ERAS-254 and trametinib
Time to achieve Cmax (Tmax) | Study Day 1 up to Day 29
  Time to achieve maximum plasma concentration of ERAS-254 and trametinib
Area under the curve (AUC) | Study Day 1 up to Day 29
  Area under the plasma concentration-time curve
Overall survival | Assessed up to 24 months from time of first dose
  Survival Status

OTHER OUTCOMES:
Duration of Response (DOR) for CNS disease in participants | Assessed up to 24 months from time of first dose
  Based on Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM)
Overall Response Rate (ORR) for CNS disease in participants | Assessed up to 24 months from time of first dose
  Based on Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM)
Disease Control Rate (DCR) for CNS disease in participants | Assessed up to 24 months from time of first dose
  Based on Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM)
Pharmacodynamic assessment | Assessed up to 24 months from time of first dose
  DUSP6: changes from baseline in the expression of DUSP-6 mRNA in blood, a marker of MAPK pathway Inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Antal, MS, Study Director — Clinical Development
Locations (29):
- United States (14):
  - University of California, San Francisco, San Francisco, California
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Florida Cancer Specialists - St. Petersburg, St. Petersburg, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Center of Nevada (CCCN), Las Vegas, Nevada
  - Oregon Health & Science University, Portland, Oregon
  - SCRI Oncology Partners (formerly Tennessee Oncology), Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - NEXT Virginia, Fairfax, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Australia (3):
  - Macquarie University, Macquarie Park, New South Wales
  - St. Vincent's Hospital, Melbourne, Victoria
  - Linear Clinical Research, LTD, Perth
- Canada (4):
  - Cross Cancer Institute- Alberta Health Services (AHS), Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - London Regional Cancer Center, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- South Korea (6):
  - Inje University Haeundae Paik Hospital, Busan, Busan Gwang'yeogsi
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital Bundang, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - The Catholic University Hospital, Seoul
- United Kingdom (2):
  - Sarah Cannon Research Institute - HCA Healthcare, City of London, London
  - Beatson West of Scotland Cancer Center, Glasgow

IPD SHARING:
Plan to Share IPD: No